CLINICAL TRIAL: NCT06757699
Title: Evaluation of Different Serum Cartilage Biomarkers in the Acute Response to Walking and Cycling in Healthy Male Subjects
Status: Available | Type: Expanded Access
Sponsor: Kocaeli University (Other)
Collaborators: Sakarya University of Applied Sciences (Unknown)
Responsible Party: Principal Investigator, Oguzhan Bahadir DEMIR, Assistant Professor, Kocaeli University
Other Study IDs: Sakarya University of Applied
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Biochemical Markers
Keywords: serum cartilage; Osteoblastic activity; Osteoclastic activity
MeSH Terms: interventions — Walking

INTERVENTIONS:
Other: Walking — Participants will perform 30 minutes of walking and cycling exercises. During the cycling and walking exercises, heart rate will be calculated using the Karvonen formula based on heart rate reserve.
  HRmax (maximum heart rate)=220-age HRR (%)(heart rate reserve)= (HR-HRrest)/(HRmax-HRrest)*100
  Blood samples will be collected from participants before starting the exercise, at the end of the 30-minute exercise session, and twice more at 30-minute intervals. The same participants will perform the cycling exercise half an hour later, and the same procedures will be applied.
Other: Cycling — Cycling

SUMMARY:
The effect of physical activity on serum cartilage biomarkers is largely unknown. This study is critical to increase our knowledge of the physiological cartilage response to activities of daily living and dynamic tasks by focusing on healthy recreationally active individuals, thus improving our understanding of the complex relationship between cartilage health and the loading that occurs during different types of loading.

DETAILED DESCRIPTION:
Biomarkers can be used to monitor cartilage metabolism and serve as prognostic or diagnostic markers to detect changes in joint structure (8). Most of these biomarkers are essential components of the cartilage extracellular matrix (ECM). The measurement of cartilage biomarkers is based on the principle that osmotic and mechanical loading triggers the efflux of proteolytically produced ECM fragments into the synovial fluid and then out of the joint capsule. Thus, biomarker concentrations can be measured by immunoassays in synovial fluid, blood, and urine. Similarly, biomarker concentrations have been used to investigate the acute or long-term effects of exercise on articular cartilage health and metabolism.

The most studied serum cartilage biomarker is cartilage oligomeric matrix protein (COMP). COMP, also known as thrombospondin-5, is a pentameric glycoprotein composed of five identical subunits. The C-terminal end of each monomer interacts with numerous KDHM proteins, such as collagen II, collagen IX, matrilins, and proteoglycans (9). In addition, COMP affects collagen secretion and fibrillogenesis, thereby influencing the rate of fibril formation, organization, and diameter (10). Due to these interactions with other KDHM proteins, COMP has an important role in the assembly and structure of the cartilage matrix, determining its mechanical properties.

Based on these properties, COMP has been widely studied in terms of acute loading and has been shown to be mechanosensitive (11). Serum COMP levels have been found to vary between -16% and +39% after 30 min of moderate running interventions (12). However, no increase in serum concentration was detected in response to other acute exercises, such as knee flexion or repeated lumbar flexion/extension (13). This suggests that the acute serum COMP response is dependent on joint loading characteristics.

Other biomarkers of interest are proteolytic enzymes involved in the degradation of cartilage KDHM components. Matrix metalloproteinases (MMPs) are a family of enzymes that vary in substrate specificity and primary structure.

Some MMP family members play a role in both KDHM remodeling and pathological degradation. For example, MMP-3 (stromelysin) degrades most components of KDHM and activates other MMPs such as MMP-9 (gelatinase B), which itself plays an important role in the development of OA (14).

YKL-40 is another KDHM protein involved in cartilage pathogenesis. Although the function of YKL-40 has not been defined in detail, it has been shown to be involved in general tissue remodeling and inflammatory processes as a glycosylase (15). YKL-40 levels increase during joint inflammation, and resistin levels are also elevated by inflammatory stimuli. Resistin is an adipokine that was initially associated with obesity and insulin resistance in rodents.

The response of MMPs, YKL-40, and resistin concentrations to exercise has been previously investigated. Marathon running has been shown to increase serum MMP-3 (+142%), YKL-40 (+56%), and resistin (+107%) concentrations immediately after the marathon compared to baseline values (16).

Type II collagen is a major component of articular cartilage. The degradation of type II collagen occurs via the activity of collagenases and MMP-9. Coll2-1 is a specific peptide epitope located on the triple helix of type II collagen molecules and is a marker of cartilage degeneration.

The nitrated form of Coll2-1 is called Coll2-1 NO2 and reflects oxidative-related cartilage matrix degradation. Serum concentrations of Coll2-1 (-13%) and Coll2-1 NO2 (-19%) have been shown to decrease after a marathon run (17).

Nagaoka et al. (18) evaluated the cartilage collagen metabolism of athletes exposed to intense joint loading. They measured both type II collagen synthesis and degradation biomarkers in urine. The results showed that type II collagen degradation increased in response to endurance exercises that included intense joint loading, especially in athletes who performed frequent jumping movements such as volleyball, basketball and handball.

The aim of our study was to examine the acute effect of two commonly used exercise interventions (walking and cycling) on the correlation of serum biomarkers reflecting cartilage extracellular matrix metabolism, COMP, YKL-40, and MMP3.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between the ages of 20-35
* Those who do physical activity for at least 30 minutes two to three days a week
* 17 healthy male individuals without any health problems will be included.

Exclusion Criteria:

* Those with acute or chronic injuries in their lower extremities
* Those with musculoskeletal disorders in their lower extremities
* Those who have undergone hip and/or knee surgery
* Those with cardio-pulmonary problems that prevent them from exercising

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healty male volunteers, physically active.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kocaeli University Faculty of Medicine Hospital, Kocaeli
  - Sakarya University Applied Sciences Physiotherapy and Rehabilitation Application and Research Center, Sakarya